CLINICAL TRIAL: NCT06756724
Title: Morphometric Insights Into Stroke Development: Analyzing Bifurcation Angles and Diameters of Common and Internal Carotid Arteries Using Frankfurt Plane Reoriented Images
Brief Title: Vessel Angles and Diameters in Stroke Disease
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Mert Nahir, Assistant professor, Tokat Gaziosmanpasa University
Other Study IDs: 22-KAEK-198
Record Dates: First submitted 2024-12-21; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Stroke Not Otherwise Specified; Control Condition
Keywords: Ischemic stroke risk; Carotid artery bifurcation; Computed tomography angiography; Bifurcation angles; Vessel diameters; Carotid artery morphology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stroke: Individuals with acute ischemic stroke
- Healthy: Individuals without any intracranial pathology

SUMMARY:
Retrospective analysis of internal carotid artery morphology on CT angiography images of patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Our study included 66 healthy individuals for control group. The control group consisted of individuals without any pathology or ischemia, selected from patients who underwent brain CTA for headache but showed no structural lesions. Additionally, none of the control group had a history of stroke or evidence of prior ischemic stroke on MRI.

Exclusion Criteria:

* After excluding patients with plaques in the carotid arteries (CCA and ICA), systemic vascular disease, risk factors for cardiogenic stroke, cardioembolism, ischemic stroke due to vasculitis or drug use, and other uncommon causes of stroke, 62 ischemic stroke patients were included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals applying to the Emergency Department of Tokat Gaziosmanpasa University Medical Faculty Hospital
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2022-09-25 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Internal carotid artery angle (degree measure) | 1 week
  The effect of angle degree change at the bifurcation point of the internal carotid artery on acute ischemic stroke
Internal carotid artery diameter (cm) | 1 Week
  Effect of internal carotid artery diameter (cm) on acute ischemic stroke.

SECONDARY OUTCOMES:
Internal carotid artery angle and diameter | 1 Week
  Statistical evaluation of the effects of changes in internal carotid artery diameter (cm) and angle (degree) on acute ischemic stroke using logistic regression analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study data may be sent for control upon request by the editor and referees. However, disclosing the data outside of publication under the relevant title may conflict with our institution's Ethics Committee principles.

REFERENCES:
- [Background] Liu Y, Ni L, Wang C, Shi P, Yin L, Fu XY, Zhou HD. Association between internal carotid artery kinking and ischemic stroke: A population-based cross-sectional study. J Stroke Cerebrovasc Dis. 2023 Dec;32(12):107417. doi: 10.1016/j.jstrokecerebrovasdis.2023.107417. Epub 2023 Nov 2. PMID 37924779
- [Background] Apaydin M, Cetinoglu K. Carotid angle in young stroke. Clin Imaging. 2021 Feb;70:10-17. doi: 10.1016/j.clinimag.2020.10.020. Epub 2020 Oct 13. PMID 33120284
- [Background] Arora S, Chien JD, Cheng SC, Chun KA, Wintermark M. Optimal carotid artery coverage for carotid plaque CT-imaging in predicting ischemic stroke. J Neuroradiol. 2010 May;37(2):98-103. doi: 10.1016/j.neurad.2009.04.002. Epub 2009 Jul 1. PMID 19573923
- [Background] Cui Y, Lv X, Wang F, Kong J, Zhao H, Ye Z, Si C, Pan L, Liu P, Wen J. Geometry of the Carotid Artery and Its Association With Pathologic Changes in a Chinese Population. Front Physiol. 2020 Jan 21;10:1628. doi: 10.3389/fphys.2019.01628. eCollection 2019. PMID 32038300